CLINICAL TRIAL: NCT05962775
Title: The Impact of Ethanol Sclerotherapy Before ART (Assisted Reproductive Technology) Cycle on Cumulative Live Birth Rate in Infertile Women With Endometrioma: A Randomized Controlled Trial
Brief Title: Ethanol Sclerotherapy Prior to ART
Acronym: START
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yavuz Emre Şükür, associate professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUTF
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Endometrioma; Infertility; Sclerotherapy; ART; IVF
Keywords: endometrioma; ethanol sclerotherapy; assisted reproductive technology; in vitro fertilization; cumulative live birth rate
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In eligible patients allocated to control group, no interventions will be done before ART cycle.
- Ethanol sclerotherapy (Experimental): In eligible patients allocated to study group, endometrioma/s will be aspirated and treated with ethanol for 10 minutes 1-2 cycles before ART.
  Interventions: Procedure: Ethanol Sclerotherapy for Endometrioma

INTERVENTIONS:
Procedure: Ethanol Sclerotherapy for Endometrioma — 2 gr IV cefazolin sodium will be administered 30 minutes before the procedure. The endometrioma cyst content will be aspirated by a single lumen needle, and the total aspirated volume calculation will be done. The endometrioma will then be washed with saline until the color of the cyst content becomes clear. Then, 96% ethanol will be injected into the cyst. The volume of injected ethanol will be 60% of the first aspirated volume (maximum 100 ml). After 10 minutes all ethanol will be aspirated.
  Arms: Ethanol sclerotherapy

SUMMARY:
The goal of this randomized controlled trial is to assess the impact of ethanol sclerotherapy on ART cycle outcomes. The main questions it aims to answer are:

1. Does ethanol sclerotherapy before ART cycle has any impact on cumulative live birth rate in patients with endometrioma?
2. Does ethanol sclerotherapy improve chronic pelvic pain, dysmenorrhea, complications during oocyte retrieval, response to ovarian stimulation (number of mature oocytes retrieved), and pregnancy loss rates?

Infertile patients with endometrioma between 4-10 cm who are scheduled for ART within 2 cycles will be randomized to ethanol sclerotherapy or no intervention.

DETAILED DESCRIPTION:
The effect of ethanol sclerotherapy before assisted reproductive technology (ART) cycle in patients with endometrioma on reproductive outcomes will be investigated. While endometrioma may result in technical difficulties in the ART process, the superiority of ethanol sclerotherapy has yet to be examined before the ART procedure in randomized controlled studies and meta-analyses. The negative effect of ethanol sclerotherapy on ovarian reserve was found to be less than other existing interventions such as cyst stripping. However, randomized controlled studies did not determine its direct effect on ART outcome. Our current study aimed to assess the effect of ethanol sclerotherapy on ART outcomes.

Infertile patients aged 18-40 years with at least one endometrioma 4-10 cm and scheduled for ART will be included in the study. Patients with any untreated thyroid dysfunction or additional disease, such as hyperprolactinemia, those who did not accept the study information and consent, and patients younger than 18 or older than 40 will not be included. Those who underwent surgery for endometrioma within 3 months before ART will be excluded. In addition, patients with an anti-mullerian hormone value below 0.3 ng/ml will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* AMH>0.3 ng/ml
* unilateral/bilateral endometrioma
* Endometrioma diameter 40-100 mm

Exclusion Criteria:

* 3 or more IVF/embryo transfer failure
* Menstrual cycle abnormalities
* Male Factor infertility
* Presence of uterine fibroids
* Presence of hydrosalpinx
* Presence of uterine abnormalities
* Suspicion of malignancy according to International Ovarian Tumor Analysis criteria

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 18 months
  live births following fresh and frozen-thaw transfer of all embryos unless pregnancy occurs

SECONDARY OUTCOMES:
pain scores | 3 months
  Visual Analog Pain Scale scores related to dysmenorrhea, dyspareunia, and/or pelvic pain will be measured before and after procedure. 0 is the lowest, 10 is the highest score. Higher the score means higher the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Batuhan Aslan, Principal Investigator — Ankara University
Locations (3):
- Turkey (Türkiye) (3):
  - Başkent University Adana IVF Center, Adana
  - Ankara University School of Medicine, Department of Obstetrics and Gynecology, Ankara
  - Bahçeci IVF Clinic, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akamatsu N, Hirai T, Masaoka H, Sekiba K, Fujita T. [Ultrasonically guided puncture of endometrial cysts--aspiration of contents and infusion of ethanol]. Nihon Sanka Fujinka Gakkai Zasshi. 1988 Feb;40(2):187-91. Japanese. PMID 3283269
- [Background] Alborzi S, Ravanbakhsh R, Parsanezhad ME, Alborzi M, Alborzi S, Dehbashi S. A comparison of follicular response of ovaries to ovulation induction after laparoscopic ovarian cystectomy or fenestration and coagulation versus normal ovaries in patients with endometrioma. Fertil Steril. 2007 Aug;88(2):507-9. doi: 10.1016/j.fertnstert.2006.11.134. Epub 2007 Apr 11. PMID 17433319
- [Background] Benaglia L, Busnelli A, Biancardi R, Vegetti W, Reschini M, Vercellini P, Somigliana E. Oocyte retrieval difficulties in women with ovarian endometriomas. Reprod Biomed Online. 2018 Jul;37(1):77-84. doi: 10.1016/j.rbmo.2018.03.020. Epub 2018 Apr 13. PMID 29759886
- [Background] Benaglia L, Somigliana E, Vercellini P, Abbiati A, Ragni G, Fedele L. Endometriotic ovarian cysts negatively affect the rate of spontaneous ovulation. Hum Reprod. 2009 Sep;24(9):2183-6. doi: 10.1093/humrep/dep202. Epub 2009 Jun 5. PMID 19502358
- [Background] Cohen A, Almog B, Tulandi T. Sclerotherapy in the management of ovarian endometrioma: systematic review and meta-analysis. Fertil Steril. 2017 Jul;108(1):117-124.e5. doi: 10.1016/j.fertnstert.2017.05.015. Epub 2017 Jun 1. PMID 28579409
- [Background] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Background] Garcia-Velasco JA, Somigliana E. Management of endometriomas in women requiring IVF: to touch or not to touch. Hum Reprod. 2009 Mar;24(3):496-501. doi: 10.1093/humrep/den398. Epub 2008 Dec 4. PMID 19056774
- [Background] Hart RJ, Hickey M, Maouris P, Buckett W. Excisional surgery versus ablative surgery for ovarian endometriomata. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004992. doi: 10.1002/14651858.CD004992.pub3. PMID 18425908
- [Background] Horton J, Sterrenburg M, Lane S, Maheshwari A, Li TC, Cheong Y. Reproductive, obstetric, and perinatal outcomes of women with adenomyosis and endometriosis: a systematic review and meta-analysis. Hum Reprod Update. 2019 Sep 11;25(5):592-632. doi: 10.1093/humupd/dmz012. PMID 31318420
- [Background] Meuleman C, Vandenabeele B, Fieuws S, Spiessens C, Timmerman D, D'Hooghe T. High prevalence of endometriosis in infertile women with normal ovulation and normospermic partners. Fertil Steril. 2009 Jul;92(1):68-74. doi: 10.1016/j.fertnstert.2008.04.056. Epub 2008 Aug 5. PMID 18684448
- [Background] Miquel L, Preaubert L, Gnisci A, Netter A, Courbiere B, Agostini A, Pivano A. Transvaginal ethanol sclerotherapy for an endometrioma in 10 steps. Fertil Steril. 2021 Jan;115(1):259-260. doi: 10.1016/j.fertnstert.2020.08.1422. Epub 2020 Oct 8. PMID 33039127
- [Background] Miquel L, Preaubert L, Gnisci A, Resseguier N, Pivano A, Perrin J, Courbiere B. Endometrioma ethanol sclerotherapy could increase IVF live birth rate in women with moderate-severe endometriosis. PLoS One. 2020 Sep 28;15(9):e0239846. doi: 10.1371/journal.pone.0239846. eCollection 2020. PMID 32986747
- [Background] Roustan A, Perrin J, Debals-Gonthier M, Paulmyer-Lacroix O, Agostini A, Courbiere B. Surgical diminished ovarian reserve after endometrioma cystectomy versus idiopathic DOR: comparison of in vitro fertilization outcome. Hum Reprod. 2015 Apr;30(4):840-7. doi: 10.1093/humrep/dev029. Epub 2015 Mar 3. PMID 25740883
- [Background] Rubod C, Jean Dit Gautier E, Yazbeck C. [Surgical management of endometrioma: Different alternatives in term of pain, fertility and recurrence. CNGOF-HAS Endometriosis Guidelines]. Gynecol Obstet Fertil Senol. 2018 Mar;46(3):278-289. doi: 10.1016/j.gofs.2018.02.013. Epub 2018 Mar 3. French. PMID 29510964
- [Background] Somigliana E, Benaglia L, Paffoni A, Busnelli A, Vigano P, Vercellini P. Risks of conservative management in women with ovarian endometriomas undergoing IVF. Hum Reprod Update. 2015 Jul-Aug;21(4):486-99. doi: 10.1093/humupd/dmv012. Epub 2015 Mar 6. PMID 25750209
- [Background] Sukur YE, Ozmen B, Yakistiran B, Atabekoglu CS, Berker B, Aytac R, Sonmezer M. Endometrioma surgery is associated with increased risk of subsequent assisted reproductive technology cycle cancellation; a retrospective cohort study. J Obstet Gynaecol. 2021 Feb;41(2):259-262. doi: 10.1080/01443615.2020.1754366. Epub 2020 Jun 4. PMID 32496142
- [Background] Yazbeck C, Madelenat P, Ayel JP, Jacquesson L, Bontoux LM, Solal P, Hazout A. Ethanol sclerotherapy: a treatment option for ovarian endometriomas before ovarian stimulation. Reprod Biomed Online. 2009 Jul;19(1):121-5. doi: 10.1016/s1472-6483(10)60055-7. PMID 19573300
- [Background] Yazbeck C, Koskas M, Cohen Scali S, Kahn V, Luton D, Madelenat P. [How I do... ethanol sclerotherapy for ovarian endometriomas]. Gynecol Obstet Fertil. 2012 Oct;40(10):620-2. doi: 10.1016/j.gyobfe.2012.07.029. Epub 2012 Sep 5. No abstract available. French. PMID 22959083